CLINICAL TRIAL: NCT03664388
Title: Registry of Patients Admitted by Acute Coronary Syndrome to University Hospital of Vigo
Brief Title: Registry of Acute Coronary Syndrome From University Hospital of Vigo
Acronym: CardioCHUVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Álvaro Cunqueiro (Other)
Responsible Party: Sponsor
Other Study IDs: Hospital Alvaro Cunqueiro
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Bleeding; Dual antiplatelet therapy
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dual antiplatelet therapy with ticagrelor/prasuglre — Compare bleeding and ischemic events according to the type and duration of dual antiplatelet therapy
  Other Names: Dual antiplatelet therapy with clopidogrel

SUMMARY:
CardoCHUVI registry was aim to study ischemic and bleeding complication after an acute coronary syndrome (ACS), both in-hospital and follow-up events.

DETAILED DESCRIPTION:
CardioCHUVI is a retrospective study aim to analyze all consecutively patients admitted by acute coronary syndrome to University Hospital Alvaro Cunqueiro of Vigo, between January 2010 to January 2018

The objective of the project was to study cardiac and bleeding complications, such as reinfarction, heart failure, atrial fibrillation, stroke, and bleeding events, together with all-cause and cardiac mortality

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to University Hospital Alvaro Cunqueiro of Vigo for acute coronary syndrome.

Exclusion Criteria:

* Secondary acute coronary syndromes during a hospital admission for another cause (i.e. acute myocardial infarction in the context of a sepsis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients admitted by acute coronary syndrome in the University Hospital Alvaro Cunqueiro of Vigo between January 2010 to January 2018
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Through study completion, an average of 3 years
  Death for any cause

SECONDARY OUTCOMES:
Reinfarction | Through study completion, an average of 3 years
  New spontaneous acute myocardial infarction
Bleeding | Through study completion, an average of 3 years
  Any bleeding according to BARC definition (from 1 to 5)
Ischemic stroke | Through study completion, an average of 3 years
  Ischemic stroke documented in CT
Cancer | Through study completion, an average of 3 years
  Any type of malignant cancer
Heart Failure | Through study completion, an average of 3 years
  Heart Failure admissions
Atrial Fibrillation | Through study completion, an average of 3 years
  Atrial fibrillation documented in ECG

CONTACTS AND LOCATIONS:
Overall Officials: Emad Abu-Assi, MD, PhD, Study Chair — University Hospital Álvaro Cunqueiro, Vigo, Spain; Sergio Raposeiras-Roubín, MD, PhD, Principal Investigator — University Hospital Álvaro Cunqueiro, Vigo, Spain; Andres Iñiguez-Romo, MD, PhD, Study Director — University Hospital Álvaro Cunqueiro, Vigo, Spain
Locations (1):
- Department of Cardiology, Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No
Registry of all consecutive patients admitted by acute coronary syndrome (ACS) to an university hospital in order to analyze bleeding and ischemic complications according to the type and duration of dual antiplatelet therapy